CLINICAL TRIAL: NCT01094418
Title: A Observational Cross Sectional Study to Evaluate the Sensory Nerve Conduction Parameters of the Distal Sensory Nerves in Patients With Impaired Glucose Tolerance and Diabetes Mellitus
Brief Title: Electrodiagnostic Parameters in Patients With Impaired Glucose Tolerance and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Geun Young Park, M.D., Ph.D.,Assistant Professor, Dept. of Rehabilitation Medicine,Bucheon St. Mary's Hospital,College of Medicine,The Catholic University of Korea
Other Study IDs: 5-2008-B0001-00099
Record Dates: First submitted 2010-03-22; First posted 2010-03-29 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Impaired Glucose Tolerance; Peripheral Polyneuropathy; DM
Keywords: polyneuropathy; Nerve conduction study; Impaired glucose tolerance test; Diabetes mellitus
MeSH Terms: conditions — Glucose Intolerance; Polyneuropathies; Diabetes Mellitus | interventions — Zinostatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IGT group: IGT diagnosed by endocrinologist
  Interventions: Other: Nerve conduction studies ( NCS) of the peripheral nerves
- DM group: DM diagnosed by endocrinologist and whose primary NCS screening shows SNAP amplitudes of sural and superficial peroneal nerves greater than 10mA DM patients with no previous diagnosis of peripheral polyneuropathy
  Interventions: Other: Nerve conduction studies ( NCS) of the peripheral nerves
- Normal healthy participants: Normal health participants with no previous history of DM, IGT, thyroid disorder, hypercholesterolemia, or other condition associated with peripheral polyneuropathy
  Interventions: Other: Nerve conduction studies ( NCS) of the peripheral nerves

INTERVENTIONS:
Other: Nerve conduction studies ( NCS) of the peripheral nerves — Standard NCS of the sural, superficial peroneal sensory nerves, peroneal, tibial motor nerves, radial and median sensory nerves, median motor nerves, F-wave studies of the Tibial and median nerves.
  NCS of the distal sensory nerves; dorsal sural Medial dorsal cutaneous and medial plantar nerves.
  Other Names: EMG(Viking )

SUMMARY:
The purpose of this study is to evaluate the distal sensory nerves of the feet, namely, the dorsal sural, medial dorsal cutaneous and medial plantar nerves, in patients with impaired glucose tolerance and diabetes mellitus type 2 and compare these parameters to those from healthy participants.

DETAILED DESCRIPTION:
Diabetic Peripheral polyneuropathy (DPP) presents as a slowly progressive primary sensory deficit in length dependent fashion, to result in the classic stocking glove distribution. There is recent evidence to indicate that patients with impaired glucose tolerance ( IGT) on OGTT, the prediabetic stage, have three times the prevalence of distal peripheral polyneuropathy than age matched controls. Patients with IGT, even in their preclinical stages, though they have less severe neuropathy than those with diabetes mellitus, have predominant sensory fiber involvement. To support this, other studies of skin biopsies of IGT patients have shown that microvascular abnormalities and neuropathic changes can occur in the prediabetic stage.

Because DPP is length dependent, it is necessary to evaluate the distal sensory nerves, other than the standard sural and superficial peroneal nerves. To support this theory, recent electrodiagnostic studies in DM patients have shown that albeit normal conduction parameters in the above mentioned two nerves, abnormal parameters can be detected in the more distal sensory nerves, such as the dorsal sural nerve, medial plantar nerves and medial dorsal cutaneous nerve.

Although the importance of evaluating the distal sensory nerves has gained much attention, no study has addressed the issue whether NCS parameters of these distal sensory nerves in IGT patients are significantly different from those of healthy controls with no medical condition, and whether these parameters are different to those with patients with diabetes mellitus, who have no previous history of peripheral polyneuropathy.

With this objective in mind, NCS of the distal sensory nerves of the feet were performed to three groups; normal healthy control group, IGT group and diabetes mellitus group.

ELIGIBILITY:
Inclusion Criteria:

* For the normal healthy control group
* Healthy participants with normal NCS parameters
* For the IGT group
* Men or women aged 20-70 with IGT referred by the department of endocrinology, with FBS 100-126 mg/dl, post 2 hour OTT - 140-200mg/dl,lasting more than one year.
* Patients willing to undergo NCS.
* For the DM group
* Men or women aged 20-70 with DM type II patients referred by the department of endocrinology, with no previous diagnosis of peripheral polyneuropathy and who showed SNAP amplitudes of the sural and superficial peroneal nerves above 10mA.
* Patients willing to undergo NCS.

Exclusion Criteria:

* No previous diagnosis of any systemic condition related to peripheral polyneuropathy (malnutrition, alcoholic hepatitis, diabetes mellitus( normal group)), no previous medication history, such as chemotherapeutics
* No symptom or sign of peripheral polyneuropathy, no history of tingling sensation, muscle weakness, or gait disturbance
* Skin lesion or swelling that would interfere with NCS conduction
* Previous diagnosis or clinical symptoms that would indicate the presence of mononeuropathy or entrapment neuropathy of the lower extremity.
* Previous trauma episode of the lower extremity
* History of alcohol ( exceeding alcohol consumption of 170g per week ) or substance abuse,
* Pregnancy
* DM group
* Presence of undiagnosed peripheral polyneuropathy determined by screening of the sural and superficial peroneal nerves.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University affiliated medical center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Nerve conduction parameters | NCS performed once, within one day after enrollment
  Nerve conduction study (NCS) parameters of the dorsal sural, medial dorsal cutaneous and medial plantar nerves, along with standard NCS of the tibial and peroenal motor, sural, superficial peronea, median and radial sensory nerves.

SECONDARY OUTCOMES:
Clinical neuropathic scoring system | once, at a single point of time, within one day after enrollment,
  The Toronoto clinical neuropathic score

CONTACTS AND LOCATIONS:
Overall Officials: Geun Young Park, MD, PhD, Principal Investigator — College of Medicine, Catholic University of Korea
Locations (1):
- Catholic University of Medicine, College of Medicine, Bucheon St. Mary's Hospital, Department of Rehabilitation Medicine, Bucheon-si, Kyoungido, South Korea